CLINICAL TRIAL: NCT03557021
Title: Impact of HIV Drug Resistance Testing, and Subsequent Change to an Individualized Therapy Based on the Resistance Profile, in Children, Adolescents and Adults With Virological Failure of Their HIV Therapy, in Three HIV Clinics in Tanzania
Brief Title: Impact of HIV Drug Resistance Testing, and Subsequent Change to an Individualized Therapy in Tanzania
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Mission Institute, Germany (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Dr. Christa Kasang, Research Coordinator, Medical Mission Institute, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIVDR2
Record Dates: First submitted 2017-09-18; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: HIV Drug Resistance

STUDY DESIGN:
Intervention Model Description: Case control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized therapy arm (Experimental): HIV Treatment failure patients will undergo an HIV Drug resistance testing and the followed therapy will be adjusted with in this setting available medications to the outcome of the resistance profile
  Interventions: Diagnostic Test: HIV Drug resistance testing
- standard therapy arm (Active Comparator): HIV Treatment failure patients will undergo an HIV Drug resistance testing and the national defined standard therapy will be applied as second line treatment.
  Interventions: Diagnostic Test: HIV Drug resistance testing

INTERVENTIONS:
Diagnostic Test: HIV Drug resistance testing — HIV Drug resistance testing by HIV pro DNA sanger sequencing

SUMMARY:
The current therapy regimens in Sub-Saharan countries, consisting of standardized first and second line drug combinations, yield a high rate of treatment failure, even within the first 12 months of therapy (23). These and other facts hint at the need for HIV resistance testing to improve treatment outcomes in resource-limited settings, but no prospective clinical data about this intervention exists. The proposed study aims to evaluate the impact of HIV drug resistance testing, and subsequent change to an individualized (second-line) therapy based on the resistance profile, in Tanzanian patients (children, adolescents and adults) with virological failure of their first-line and second-line therapy. Additionally, prevalence, patterns and clinical impact of HIVDR will be assessed, as well as the effect of enhanced adherence counselling.

The results of this study will help doctors to take evidence-based diagnostic and therapeutic decisions at an individual level, and will inform policy-makers in their decisions about future treatment and management concepts for HIV/AIDS.

DETAILED DESCRIPTION:
HIV/AIDS is one of the main health challenges of our time, with a global burden of disease higher than any other infectious disease. The widespread use of antiretroviral drugs has changed its face from a fatal fate to a chronic disease. However, there are still many differences in the standard of care globally. Drug resistance testing is routinely performed in high income countries, but is often not available in resource limited settings. Instead, treatment consists of standardized therapy regimes, chosen from a limited amount of antiretroviral drugs. This may contribute to the high rates of virological failure seen in patients, and especially children and adolescents, on therapy. Virological failure persisting despite intensified enhanced adherence-counselling result in poor treatment success in HIV infected adults, children and adolescents on treatment and therefore early deaths. If therapy failure occurs, and HIV drug resistance is the likely reason, physician in Tanzania need to blindly choose a second-line therapy regimen, without knowledge of the exact resistance profile. However, multiple studies have discovered high rates of HIV drug resistance in patients with first line treatment failure, and even in therapy-naïve patients. To obtain information about presence of resistance mutations HIV genotypic resistance testing is required. This test is used to detect HIV genomic mutations that confer resistance to specific types of antiretroviral drugs as an aid in monitoring and treating HIV-infection. The test identifies mutation on the protease and reverse transcriptase gene, which are responsible for very crucial steps in the viral replication process. Results from this test can identify the medication for whom the virus is still susceptible and for whom it is already resistant. With this, it can be avoid switching to second-line regimen without the knowledge of the presence or absence of antiretroviral drug resistance. An individualized therapy can follow making sure that medication works best and the clinical outcome can increase.

While the positive impact of HIV resistance testing on treatment outcomes in high-income countries is well established, no prospective data has been published about the effect in resource-limited settings. This absence of data poses a hole in clinical knowledge, because the results from high-income countries are not readily transferable to low-income settings.

The proposed study aims to evaluate the impact of HIV drug resistance testing, and subsequent change to an individualized (second-line) therapy based on the resistance profile, compared to standardized second-line therapy. The study is designed as a randomised controlled trial. The study participants, Tanzanian patients (children, adolescents and adults) with virological failure of their first-line therapy, will be recruited at several study sites. All patients will first receive enhanced adherence counselling. The patients that still show virological failure three months after the counselling will be eligible for resistance testing. The regimen will be switched to individualized (second-line) ART or standardized second-line ART, and clinical, immunological and virological outcome parameters will be collected in a 6 month and 12 month follow up visit (Group I,II,III IV). In addition to the outcome of individualized therapy, the proposed study would yield insights about the prevalence and patterns of HIV drug resistance in patients with failure of their first-line therapy, and also about the effectiveness of enhanced adherence counselling.

For ethical reasons also 250 seconnd line treatment failure patients (Group V) with fast clinical progress will be included and transfered directly to the individualized therapy arm. With that we hope to bring them back to a working treatment.

The main diagnostic method of this study, HIV genomic sequencing, will be implemented and performed at the National Institute for Medical Research in Mwanza, Tanzania. This will contribute directly to the HIV-related diagnostic capacities of Tanzanian laboratories.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV positive patients on first-line ART
2. Virological treatment failure with > 1000 copies/ ml

Exclusion Criteria:

1. No consent given
2. HIV patients with psychiatric disorders

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Viral Load | 12 month
  Viral load will be measured by plasma HIV viral load measurement (copies per ml) after switching first-line treatment failure patients to individualized therapy compared to standard second line therapy.

SECONDARY OUTCOMES:
Incidence of HIV related adverse events at 6 month | 6 month
  HIV related adverse events at 6 month will be determined according to CTC AE list version 4
Incidence of HIV related adverse events at at 12 month | 12 month
  HIV related adverse events at 6 month will be determined according to CTC AE list version 4
Prevalence of HIV Drug resistance mutations | study start
  The prevalence of HIV drug resistance mutations will be determined in patients with virological failure of first-line antiretroviral therapy
Pattern of HIV Drug resistance mutations | study start
  The patterns of HIV drug resistance mutations will be determined in patients with virological failure of first-line antiretroviral therapy
Viral load at 3th month | 3 month
  Viral load will be measured by plasma HIV viral load measurement (copies per ml) after enhanced conselling.

CONTACTS AND LOCATIONS:
Overall Officials: John Changalucha, MD, Study Chair — National Institute of Medical research Mwanza
Locations (3):
- Tanzania (3):
  - PASADA, Dar es Salaam
  - Baylor Hospital, Mwanza
  - Bugando Medical Center, Mwanza

IPD SHARING:
Plan to Share IPD: Undecided